CLINICAL TRIAL: NCT01797913
Title: The Study of Gemcitabine in the Maintenance Treatment of Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, Vice director of department of chemotherapy, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-CJH
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: THE Efficacy and Safety of Gemcitabine in the Maintenance Treatment of Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — Gemcitabine

ARMS (1):
- gemcitabine (Experimental)
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: gemcitabine — gemcitabine，1000mg/m2，ivgtt，DAY1&DAY8

SUMMARY:
assess the efficacy and safety of gemcitabine in the maintenance treatment of advanced non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

18~75 years Patients who were diagnosed by the histologic, cytologic diagnosis of IIIb-IV non-small cell lung cancer patients who have acceptted combination chemotherapy based on platinum 4 course,SD OR PR,the CR patients should accept 6 course of combination chemotherapy.

3~8 weeks after patients complete first line chemotherapy(include radiotherapy) Ecog0-2 Expected life time longer than 3 monthes

Normal laboratory values:

* leucocyte ≥ 4×109/L
* neutrophil ≥ 1.5×109/L
* platelet ≥ 100×109/L
* Hemoglobin ≥ 10g/L
* ALT and
* AST ≤ 2.5×ULN (≤ 5×ULN if liver metastasis) Signed written informed consent

Exclusion Criteria:

* Patients have used drugs according to protocol
* Uncontrolled infection of Bacterial or virus or fungal
* Patients with other malignant tumor
* Uncontrolled brain metastases
* Female patients during their pregnant and lactation period, or patients without contracep

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-08; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
PFS | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China